CLINICAL TRIAL: NCT06281912
Title: Impact of Anti PD-1 Therapy in Children, Adolescents and Young Adults (CAYA) Melanoma Patients
Acronym: MELCAYA
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Perugia (Other)
Responsible Party: Principal Investigator, Mario Mandalà, Associate Professor, Azienda Ospedaliera di Perugia
Other Study IDs: 4504/23
Record Dates: First submitted 2023-09-22; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Early Melanoma; Advanced Melanoma
Keywords: PD-1 antibodies, childhood, adolescent, melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adolescent/childhood: patients <20 years old with with stage III and IV melanoma diagnosis
- young adult: patients < 30 years with stage III and IV melanoma diagnosis

SUMMARY:
This is a retrospective observational cohort study, the primary objective is investigate the activity and efficacy of anti PD-1 antibodies in children, adolescents and young adult melanoma patients, with radically resected or metastatic disease

DETAILED DESCRIPTION:
The aim of the study is to evaluate the activity and efficacy of anti PD-1 antibodies in adolescent, childhood and young adult with early and advanced melanomas through a multicenter transnational European retrospective analysis Clinical outcomes will be retrospectively retrieved beginning from the primary diagnosis of melanoma. Clinical outcomes will be retrospectively evaluated starting from the time of start of treatment for up to a the most recent follow-up. Data collected will include demographic information, disease history, baseline conditions, clinical outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged ≥ 12 years;
2. Histologically confirmed melanoma;
3. Anti PD-1 Immunotherapy (Ipilimumab plus Nivolumab);
4. Previous and subsequent treatments will be collected;
5. Clinical and follow-up data available

Exclusion Criteria:

1. No immunotherapy received;
2. No melanoma;
3. Age > 30 yrs

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent, childhood and young adult with early and advanced melanomas treated with anti PD-1 therapy
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
rate of objective response | 12 months
  efficay of anti PD-1 antibodies in adolescent, childhood and young through Tumor assessment revision adult with early and advanced melanomas

SECONDARY OUTCOMES:
adverse event incidence | 12 months
  Number of AE occurred during treatment defined using CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (13):
- France (2):
  - Aix-Marseille Universite, Marseille
  - Institut Curie, Paris
- Germany (3):
  - Ospedale universitario della Charité, Berlin
  - German Cancer Research Center (Deutsches Krebsforschungszentrum (DKFZ), Heidelberg
  - University Children's Hospital Tuebingen, Tübingen
- Italy (3):
  - Universita Degli Studi Di Firenze, Florence
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Universita Cattolica Del Sacro Cuore, Roma
- Princess Máxima Center for Pediatric Oncology (Prinses Máxima Centrum voor kinderoncologie), Utrecht, Netherlands
- Narodowy Instytut Onkologii Im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw, Poland
- Spain (2):
  - Institut Catala D'Oncologia, Barcelona
  - Instituto de Investigaciones Biomédicas August Pi i Sunyer, Barcelona
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No